CLINICAL TRIAL: NCT03658291
Title: Sanjin Tablets for the Treatment of Acute Simple Lower Urinary Tract Infection and Its Influence on Recurrence Rate: a Randomized, Double Blind, Parallel Control of Positive Drugs, Multi-center Clinical Study
Brief Title: Clinical Study of Sanjin Tablets for the Treatment of Acute Simple Lower Urinary Tract Infection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Academy of Chinese Medical Sciences (Other)
Collaborators: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other); Shanghai University of Traditional Chinese Medicine (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Hubei Hospital of Traditional Chinese Medicine (Other); Chengdu University of Traditional Chinese Medicine (Other); Yunnan Provinical Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Yanming Xie, Deputy director, China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Sanjin tablets
Record Dates: First submitted 2018-07-24; First posted 2018-09-05 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Urinary Tract Infection Lower Acute
Keywords: Sanjin tablets; efficacy and safety; recurrence rate; randomized; double blind; parallel control; multi-center clinical study
MeSH Terms: interventions — Levofloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sanjin tablets group (Experimental): Sanjin tablets+ levofloxacin simulants
  Interventions: Drug: Sanjin tablets
- Levofloxacin group (Placebo Comparator): Sanjin tablets simulants +levofloxacin
  Interventions: Drug: Sanjin tablets simulants
- Sanjin tablets+ Levofloxacin group (Active Comparator): Sanjin tablets+ levofloxacin
  Interventions: Drug: Levofloxacin

INTERVENTIONS:
Drug: Sanjin tablets — Sanjin tablets,3 pills /time, 4 times/ day, for 7 days+levofloxacin simulants,0.1g, po bid, for 7 days.
  Other Names: levofloxacin simulants
  Arms: Sanjin tablets group
Drug: Sanjin tablets simulants — levofloxacin ,0.1g, po bid, for 7 days+Sanjin tablets simulants,3 pills /time, 4 times/ day, for 7 days.
  Other Names: Levofloxacin
  Arms: Levofloxacin group
Drug: Levofloxacin — Sanjin tablets,3 pills /time, 4 times/ day, for 7 days+levofloxacin,0.1g, po bid, for 7 days.
  Other Names: Sanjin tablets
  Arms: Sanjin tablets+ Levofloxacin group

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and immune mechanism of Sanjin tablets for the treatment of acute simple lower urinary tract infection and its influence on recurrence rate.

DETAILED DESCRIPTION:
In order to evaluating the efficacy, safety and immune mechanism of Sanjin tablets for the treatment of acute simple lower urinary tract infection and its influence on recurrence rate and through research data to guide clinical, improving the rational use of drugs, especially the rational application of antibiotics. In this study, a randomized, double blind, parallel control of positive drugs, multi-center clinical study will be established. According to the relevant regulations of the CFDA, 252 cases need to be registered at least. These cases will be divided into treatment group（Sanjin tablets+ levofloxacin simulants），control group 1（Sanjin tablets simulants +levofloxacin）and control group 2（Sanjin tablets+ levofloxacin）. Each group will be treated for 7 days and followed up for 2 times. The efficacy indicators of this study were mainly from three dimensions: syndrome, laboratory routine examination and bacteriology examination. The symptom scores and cytokine changes of each group before and after treatment were observed.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 18 to 50 years of age.
2. Meets the western diagnostic criteria of acute simple lower urinary tract infection, the disease duration does not exceed 72 hours.
3. Urine retention in the screening period -1-0 days, bacterial culture results were sensitive to levofloxacin.(Urine retention for bacterial culture and clinical treatment at the same time)
4. The syndrome differentiation of TCM is syndrome of dampness-heat in lower jiao.
5. Did not receive antibiotic treatment within 48 hours Before being selected.
6. The inclusion of those who confirmed not pregnant
7. Those who agree to participate in this clinical trial and sign the informed consent, the process of informed consent meet the relevant provisions of the GCP.

Exclusion Criteria:

1. Those who are allergic to the test drug ingredients or quinolones.
2. In the past, there was a history of bacterial culture that was not sensitive to levofloxacin.
3. Diagnosed as complicated urinary tract infection.
4. Patients with urinary calculi or obstruction, urinary tuberculosis, renal papillary necrosis, perinephric abscess or neurogenic bladder.
5. Combined with vaginitis symptoms, genital ulcers or gonorrhea.
6. Combined with severe cardiopulmonary disease, liver and kidney disease, advanced tumor, blood, central nervous system (such as the history of epilepsy) or other serious or progressive disease.
7. A patient who has a neurological or mental illness and cannot cooperate.
8. Infected persons who must use other antibacterial drugs in combination.
9. Pregnancy, lactating women or recent birth planners.
10. Those who have participated in other clinical trials within 3 months before being selected.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 252 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
The lower urinary tract infection symptoms of 252 participants will be assessed | After 7 days of medication
  The symptoms mainly includes frequent urination,urgent urination,urinary pain, lower abdominal pain and pain in the kidney area.If these symptoms disappear after 7 days of medication,it indicates the subject is cured.

SECONDARY OUTCOMES:
The urine leukocyte of 252 participants will be assessed | After 7 days of medication
  If the urine leukocyte return to normal value after 7 days of medication,it indicates the subject is cured.
The bacteriological examination of 252 participants | After 7 days of medication
  If the original infected part of the specimen did not regenerate the original infected pathogen after 7 days of medication,it indicates the subject is cured.
The recurrence rate of subjects who is cured in 252 participants will be assessed by lower urinary tract infection symptoms | 28 days after the end of treatment
  If the lower urinary tract infection symptoms of subjects who is cured appears again in the fourth week after end of medication,it indicates the subject has relapsed.
The recurrence rate of subjects who is cured in 252 participants will be assessed by urine leukocyte | 28 days after the end of treatment
  If the urine leukocyte value of subjects who is cured rises again in the fourth week after end of medication,it indicates the subject has relapsed.
The recurrence rate of subjects who is cured in 252 participants will be assessed by bacteriological examination | 28 days after the end of treatment
  If the urine culture of subjects who is cured indicates that the original urinary tract pathogen is positive again in the fourth week after end of medication,it indicates the subject has relapsed.

CONTACTS AND LOCATIONS:
Overall Officials: Yanming Xie, BA, Principal Investigator — Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lyu J, Xie YM, Gao Z, Shen JW, Deng YY, Xiang ST, Gao WX, Zeng WT, Zhang CH, Yi DH, Wang LX, Wang ZF. Sanjin tablets for acute uncomplicated lower urinary tract infection (syndrome of dampness-heat in the lower jiao): protocol for randomized, double-blind, double-dummy, parallel control of positive drug, multicenter clinical trial. Trials. 2019 Jul 19;20(1):446. doi: 10.1186/s13063-019-3539-5. PMID 31324199